CLINICAL TRIAL: NCT07205822
Title: A Phase IIIb, Open-label, Multinational Study Assessing the Efficacy and Safety of Dato-DXd Treatment in Patients With HRpositive, HER2 IHC 0, Locally Advanced Inoperable or Metastatic Breast Cancer Refractory to Endocrine Therapy (TROPION-Breast06)
Brief Title: A Study of Dato-DXd in Inoperable or Metastatic Hormone Receptor-positive, HER2 IHC 0 Breast Cancer
Acronym: TB06
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9260C00003; 2025-521904-23-00 (Other: CTIS (EU))
Record Dates: First submitted 2025-09-11; First posted 2025-10-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: HR+, HER2 IHC 0, LA Inoperable/Metastatic, Endo Refractory
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm group (Experimental): All participants will receive Dato-DXd (6 mg/kg IV on Day 1, Q3W; up to a maximum of 540 mg Q3W for participants ≥ 90 kg) until investigator-defined disease progression according to RECIST 1.1 or until unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met.
  Interventions: Drug: Dato-DXd

INTERVENTIONS:
Drug: Dato-DXd — All participants will receive Dato-DXd (6 mg/kg IV on Day 1, Q3W; up to a maximum of 540 mg Q3W for participants ≥ 90 kg) until investigator-defined disease progression according to RECIST 1.1 or until unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met. Continued treatment with the same study drug post-progression may be allowed, based on prior discussion with sponsor/sponsor representative/study physician on a case-by-case basis following written investigator's confirmation of continuing clinical benefit to the patient post progression. The study is anticipated to enrol for an 18-month period, and DCO is expected to occur approximately 6 months after the last participant has been dosed.
  Other Names: IMP administration

SUMMARY:
A study to assess the efficacy and safety of Dato-DXd in the pre-chemotherapy setting for patients with metastatic HR-positive, HER2 IHC 0 breast cancer.

DETAILED DESCRIPTION:
This is a Phase IIIb, single-arm, open-label, multicentre, multinational study assessing the efficacy and safety of Dato-DXd in participants with HR-positive, HER2 IHC 0, locally advanced inoperable or metastatic breast cancer refractory to endocrine therapy.

Refer to the study schema (Figure 1) and SoA (Section 1.3) for overall design and required assessments. Day 1 is defined as the first day of study treatment.

Approximately 100 participants will be treated in this study with Dato-DXd 6 mg/kg as an intravenous infusion every 3 weeks (21-day cycle), up to a maximum of 540 mg for patients ≥ 90kg. Participants will receive study intervention until RECIST 1.1 defined radiological progression by investigator unless there is evidence of unacceptable toxicity or if the participant requests to stop the study treatment.

Written consent is required from all participants for newly acquired tumour biopsy collection at baseline or for providing a tumour biopsy sample collected within 6 weeks prior to initiating Dato-DXd and, if feasible, at progression. This sample will be used to assess for HER2 and TROP2 expression and exploratory analysis of biomarkers of response. Participants are also expected to consent for repeated liquid biopsy at baseline, during the treatment period, and at progression to evaluate biomarkers of response and resistance. (Sample collection in China will comply with local regulatory requirements.) Tumour imaging will occur every 8 weeks (± 1 week) after the first dose of study drug for 48 weeks and then every 12 weeks (± 1 week) thereafter until RECIST 1.1 disease progression as assessed by the investigator or the start of subsequent anticancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years (and above legal age) at the time of screening.
2. Inoperable or metastatic HR-positive, HER2 IHC 0 breast cancer (per ASCO/CAP guidelines, on local laboratory results); ie, is documented as HR-positive (either ER and/or PgR positive [ER or PgR ≥ 1%]) and HER2 IHC 0 (defined as no staining or incomplete and faint/barely perceptible membrane staining in ≤ 10% of tumour cells).
3. Progressed on and not suitable for further endocrine therapy per investigator assessment.
4. ECOG performance status of 0 or 1, with no deterioration over the previous 2 weeks prior to the first dose of study intervention.
5. Minimum life expectancy of 12 weeks at screening.
6. Provision of acceptable tumour sample (no more than 6 weeks old) prior to the first dose of study intervention or retrospectively as defined in the Laboratory Manual and the Diagnostic Testing Manual
7. Participants must have measurable disease as per RECIST 1.1 or evaluable disease. Lesions that will be subject to mandatory biopsy before, during, and after the dosing cannot be considered as TLs as per RECIST requirements.
8. Adequate bone marrow reserve and organ function within 7 days before the first dose of study intervention.

   1. Haemoglobin ≥ 9.0 g/dL (red blood cell/plasma transfusion is not allowed within 1 week prior to screening assessment).
   2. Absolute neutrophil count ≥ 1.5×109/L (granulocyte colony stimulating factor administration is not allowed within 1 week prior to screening assessment).
   3. Platelet count ≥ 100×109/L (platelet transfusion is not allowed within 1 week prior to screening assessment).
   4. Serum albumin ≥ 2.5 g/dL.
   5. TBL ≤ 1.5 × ULN or ≤ 3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinaemia).
   6. Except in the setting of HBV, ALT and AST ≤ 2.5 × ULN; for participants with hepatic metastases, ALT and AST ≤ 5 × ULN. See Exclusion Criterion 8 for requirements in the setting of HBV.
   7. Calculated CrCL ≥ 30 mL/min as determined by Cockcroft Gault (using actual body weight).
9. Male and/or female assigned at birth, inclusive of all gender identities.
10. Contraceptive use by participants or participant partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies;

    (a) Male participants: (i) Use of a condom plus an additional contraceptive method, or avoid intercourse from enrolment and throughout study for at least 4 months after the last dose of Dato-DXd, in addition to the female partner using a highly effective contraceptive method.

    (ii) Starting at the time of first dose of Dato-DXd, male participants must not freeze or donate sperm at any time during this study and for at least 4 months after the last dose of Dato-DXd. Preservation of sperm should be considered prior to the first dose of study intervention.

    (b) Female participants:Female participants not of child-bearing potential (ii) Female participants receiving HRT and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for WOCBP if they wish to continue using HRT during the study. Otherwise, HRT must be discontinued to allow confirmation of post-menopausal status prior to study enrolment; (iii) WOCBP must use one highly effective form of contraception or avoid intercourse from enrolment throughout study and for at least 7 months after the last dose of Dato-DXd. All WOCBP must have a negative serum pregnancy test documented during screening.

    (iv) Starting at the time of first dose of Dato-DXd, female participants must not donate, or retrieve for their own use, ova at any time during this study and for at least 7 months after the last dose of Dato-DXd. Preservation of ova should be considered prior to the first dose of study intervention.
11. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this CSP.
12. All races, genders, and ethnic groups are eligible for this study.

Exclusion Criteria:

1. As judged by the investigator, any evidence of diseases (such as severe or uncontrolled systemic diseases, including active bleeding diseases and significant cardiac or psychological conditions), history of allogenic organ transplant, and/or substance abuse which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol.
2. History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non melanoma skin cancer (basal cell carcinoma of the skin or squamous cell carcinoma of the skin) and curatively treated in situ disease.
3. Persistent toxicities caused by previous anticancer therapy, excluding alopecia, not yet improved to Grade ≤ 1 or baseline. Note: participants may be enrolled with some chronic, stable Grade 2 toxicities (defined as no worsening to Grade > 2 for at least 3 months prior to the first dose of study intervention and managed with SoC treatment) which the investigator deems related to previous anticancer therapy):

   1. Chemotherapy-induced neuropathy
   2. Fatigue
   3. Residual toxicities from prior immunotherapy treatment: Grade 1 or Grade 2 endocrinopathies, which may include but are not limited to hypothyroidism/hyperthyroidism, Type I diabetes, hyperglycaemia, adrenal insufficiency, or adrenalitis; and skin hypopigmentation (vitiligo) Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention in the opinion of the investigator may be included (eg, hearing loss).
4. Spinal cord compression or brain metastases (unless asymptomatic, stable, and not requiring treatment with corticosteroids or anticonvulsants for at least 2 weeks prior to the first dose of study intervention). Participants with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants must have recovered from the acute toxic effect of radiotherapy (eg, dizziness and signs of increased intracranial pressure). A minimum of 2 weeks must have elapsed between the end of brain radiotherapy and the first dose of study intervention. A minimum of 3 days must have elapsed between the end of corticosteroid therapy for CNS metastatic disease and the first dose of study intervention.
5. Leptomeningeal carcinomatosis or metastasis.
6. Has significant third-space fluid retention (eg, ascites or pleural effusion) and is not amenable for required repeated drainage.
7. Clinically significant corneal disease.
8. Has active or uncontrolled hepatitis B or C virus infection. Participants are eligible if they:

   1. Have been curatively treated for HCV infection as demonstrated clinically and by viral serologies
   2. Have received HBV vaccination with only anti-HBs positivity and no clinical signs of hepatitis
   3. Are HBsAg- and anti-HBc+ (ie, those who have cleared HBV after infection) and meet conditions i-iii of criterion 'd' below:
   4. Are HBsAg+ with chronic HBV infection (lasting 6 months or longer) and meet conditions i-iii below:

   (i) HBV DNA viral load < 2000 IU/mL (ii) Have normal transaminase values or, if liver metastases are present, abnormal transaminases, with a result of AST/ALT < 3 × ULN, which are not attributable to HBV infection (iii) Start or maintain antiviral treatment if clinically indicated as per the investigator
9. Known HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA, CD4+ count ≥ 350, no history of AIDS defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen). If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4+ count is recommended. Participants must be tested for HIV during the screening period if acceptable by local regulations or an IRB/EC.
10. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals; suspected infections (eg, prodromal symptoms); or inability to rule out infections (participants with localised fungal infections of skin or nails are eligible).
11. Known to have active tuberculosis infection (clinical evaluation that may include clinical history, physical examination, and radiographic findings, or tuberculosis testing in line with local practice).
12. Resting ECG with clinically abnormal findings.
13. Uncontrolled or significant cardiac disease including:

    1. Myocardial infarction or uncontrolled/unstable angina within 6 months before the first dose of study intervention.
    2. Congestive heart failure (New York Heart Association Class II to IV).
    3. Uncontrolled hypertension (resting systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg).
    4. Cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (NCI CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted based on the investigator judgement with cardiologist consultation recommended.
14. History of non-infectious ILD/pneumonitis, including radiation pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
15. Has severe pulmonary function compromise.
16. Prior exposure to the following anticancer therapies:

    1. Any TROP2-targeted therapy.
    2. Any treatment (including ADC) containing a chemotherapeutic agent targeting topoisomerase I.
    3. Any chemotherapy in the metastatic setting.
17. Prior exposure to chloroquine/hydroxychloroquine without an adequate treatment washout period of > 14 days before the first dose of study intervention.
18. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, tumour embolisation, or monoclonal antibodies ≤ 3 weeks [for small molecule targeted agents: ≤ 2 weeks or 5 half-lives, whichever is longer, prior to the first dose of study intervention]). Herbal or natural products intended as treatment or prophylaxis for any type of cancer that may interfere with the activity of the study intervention are excluded.
19. Any concurrent anticancer treatment with the exception of bisphosphonates, denosumab for the treatment of bone metastases.

    Concurrent use of hormonal therapy for non cancer related conditions (eg, HRT) is allowed.
20. Received prior radiotherapy to the chest within 4 weeks of the start of study intervention or has ongoing radiation-related toxicities requiring corticosteroids.
21. Palliative radiotherapy with a limited field of radiation within ≤ 2 weeks or with wide field of radiation to chest or to more than 30% of the bone marrow within ≤ 4 weeks prior to the first dose of study intervention.
22. Curative radiotherapy; however, palliative radiotherapy for optimal symptom control or pain management is allowed.
23. Concomitant use of chronic systemic (IV or oral) corticosteroids or other immunosuppressive medications > 10 mg/day of prednisone or equivalent, except for managing AEs; inhaled steroids, intra-articular steroid injections, and other topical steroid formulations are permitted in this study.
24. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within ≤ 3 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
25. Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 4 weeks (unless the safety profile is known prior to the first dose of study intervention), enrolment into a prior Dato-DXd study regardless of treatment assignment, or concurrent enrolment in another clinical study (unless the study is observational [non-interventional], or the participant is in the follow-up period of an interventional study).
26. Participants with a known history of severe hypersensitivity reactions to either the drug or inactive excipients (including but not limited to polysorbate 80) of Dato-DXd.
27. Participants with a known history of severe hypersensitivity reactions to other monoclonal antibodies.
28. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
29. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
30. Previous enrolment in the present study.
31. For females only: is pregnant (confirmed with positive serum pregnancy test) or breastfeeding or planning to become pregnant.
32. Female participants should refrain from breastfeeding from enrolment throughout the study and for at least 7 months after last dose of study intervention.
33. Participants for whom the use of steroid-containing mouthwash in contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-02-02 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per RECIST 1.1 as assessed by the investigator | From date of first dose of study intervention until disease progression per RECIST 1.1 or death from any cause, whichever occurs first, assessed up to approximately 24 months
  PFS is defined as time from date of first dose of study intervention until progression per RECIST 1.1 as assessed by the investigator or death due to any cause.

SECONDARY OUTCOMES:
Proportion of participants with oral mucositis/stomatitis | From date of first dose of study intervention until 28 days after the last dose (Safety Follow-up)
  Proportion of participants with oral mucositis/stomatitis
Proportion of participants with ocular events | From date of first dose of study intervention until 28 days after the last dose (Safety Follow-up)
  Proportion of participants with ocular events
Proportion of participants with Grade 3 or higher Adverse Events (AEs) possibly related to Dato-DXd treatment | From date of first dose of study intervention until 28 days after the last dose (Safety Follow-up)
  Grade 3 or higher adverse events possibly related to Dato-DXd treatment (Grade ≥ 3 treatment-related adverse events) according to NCI CTCAE 5.0. Possibly related is defined as reasonable possibility that the adverse event was caused by investigational product, as assessed by investigator. Missing responses are counted as possibly related.
Clinical benefit rate (CBR) at 24 weeks | At 24 weeks after first dose
  CBR at 24 weeks is defined as the percentage of participants who have a confirmed CR or PR or who have SD per RECIST 1.1 as assessed by the investigator and derived from the raw tumour data for at least 24 weeks after date of first dose.
Objective response rate (ORR) | From date of first dose until disease progression or death, whichever occurs first, assessed up to approximately 24 months
  ORR is defined as the proportion of participants with measurable disease at baseline who have a confirmed CR or confirmed PR, as assessed by the investigator and derived from raw tumour data per RECIST 1.1.
Duration of response (DoR) | From the date of first documented confirmed response until disease progression per RECIST 1.1 or death from any cause, whichever occurs first, assessed up to approximately 24 months
  DoR will be defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 as assessed by the investigator or death due to any cause. The analysis will include all dosed participants who have a confirmed response.
Overall survival (OS) | From date of first dose of study intervention until death from any cause, assessed up to approximately 24-30 months
  OS defined as the time from the date of the first dose of study intervention until the date of death due to any cause. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy

CONTACTS AND LOCATIONS:
Locations (33):
- United States (6):
  - Research Site, Largo, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Houston, Texas
  - Research Site, Puyallup, Washington
- China (7):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Linyi
  - Research Site, Shandong
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- France (5):
  - Research Site, Clermont-Ferrand
  - Research Site, La Roche-sur-Yon
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pierre-Bénite
- Italy (6):
  - Research Site, Aviano
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
- South Korea (3):
  - Research Site, Bukgu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/